CLINICAL TRIAL: NCT06061822
Title: Artificial Intelligence Delivered Cardiac Magnetic Resonance - Prospective Validation
Acronym: AID-MR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other); Medical Research Council (Other Government); Rosetrees Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 23HH8238
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Healthy Volunteers
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-planned images acquired (Experimental)
  Interventions: Diagnostic Test: AI-assisted cardiac magnetic resonance imaging
- Radiographer-planned images acquired (Active Comparator)
  Interventions: Diagnostic Test: AI-assisted cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: AI-assisted cardiac magnetic resonance imaging — An AI algorithm will be used to automatically position (plan) the scan planes used in a cardiac MRI scan. The resultant images will be compared with standard radiographer-positioned images.

SUMMARY:
Cardiac MRI (CMR) scanning allows doctors to create detailed images of the heart. However, the need for experienced cardiac radiographers to perform each scan can make CMR's delivery difficult, and some patients in the UK wait more than half a year for a scan. These radiographers must take pictures of different part of the heart, termed "views", each of which must be precisely positioned.

The investigators believe they can revolutionise CMR, by using artificial intelligence to automatically position the views so radiographers can focus on more difficult tasks.

The investigators have used a retrospective database of pseudonymised (anonymised and linked) CMR scans at our hospital to create these artificial intelligence (AI) algorithms, and they have validated them retrospectively on previous studies. The investigators now wish to test the algorithms prospectively.

In this study, the investigators will recruit patients undergoing clinical CMR scans. In addition to the routine images acquired by expert radiographers, the investigators will require a duplicate set of images, positioned and planned by the AI algorithms.

The investigators will then compare, within each patient, the AI-planned and expert-radiographer-planned scanning in terms of both speed and image quality.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged at least 18 years)

Exclusion Criteria:

* Children (patients below age 18).
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Time taken to acquire images | During the MRI scan
  The time taken in seconds from the beginning of the planning process, until the last planned images has been fully acquired.
Image quality | During the MRI scan
  Quality of acquired images (AI-planning versus radiographer planning) assessed by level 3 cardiac MRI accredited doctors, by asking them to choose whether (a) the AI-acquired image is of higher diagnostic quality, (b) the radiographer-acquired image is of higher diagnostic quality, or (c) the AI- and radiographer-acquired images are of identical diagnostic quality.

CONTACTS AND LOCATIONS:
Overall Officials: James P Howard, MB BChir PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We are considering consenting patients to have their IPD shared. This would comprise anonymised images from the scan, with the AI-acquired and radiographer-acquired images indicated as such.